CLINICAL TRIAL: NCT00845247
Title: The Effect of Case Management in Complex Cancer Pathways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other); The Research Council for Health and Disease, Denmark (Other); Danish Cancer Society (Other); Novo Nordisk A/S (Industry); Kvalitets- og efteruddannelsesudvalget for Region Midtjylland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 477 980 567; Datatilsyn J.nr. 2008-41-2932
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Colonic Neoplasms; Rectal Neoplasms
Keywords: Case Management
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Control group patients will receive usual medical plus usual supportive treatment.
- Case management (Active Comparator): Intervention group patients are offered the support of a nurse case manager throughout their course of treatment.
  Interventions: Other: Nurse case management

INTERVENTIONS:
Other: Nurse case management — Intervention group patients are offered the support of a nurse case manager throughout their course of treatment.
  Arms: Case management

SUMMARY:
Introduction: Case management (CM) has been proposed as a method for optimizing the course of treatment for complicated cancer patients. However evidence of the effect of CM is limited and methodologically rigorous research is needed.

Aim: To analyze effects of Nurse CM in complicated cancer care.

Methods: The study is designed as a two-arm randomized controlled trial (RCT) including approximately 280 colorectal cancer patients.

Intervention group patients will be offered usual medical treatment plus supportive intervention from a case manager. Control group patients will receive usual medical and supportive treatment.

The intervention: Case managers are registered nurses and possess thorough knowledge of cancer treatment and pathways. Core intervention elements: Planned and ad hoc personal and telephone contacts, surveillance of care pathways, coordination and dissemination of care plan (including transfer of patient-specific information to other departments and general practice).

Primary outcomes: Patient evaluations of care pathways and "Quality of Life" (questionnaires).

Secondary outcomes: Use of health care services and care process measures (The National Health Insurance Service Registry and The National Patient Registry; and GPs' evaluations of continuity of care (questionnaire).

Schedule:

* "Case management used to optimize cancer care pathways: A systematic Review" has been published in BMC Health Services Research.
* The CM manual has been written. Questionnaires are under development and pilot testing.
* Two case managers have been appointed 1. January 2009.
* After training and pilot testing of the intervention the RCT will begin in March 2009. Inclusion period is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal cancer are highly suspected and a course of treatment at Department P, Aarhus University Hospital is expected to follow.

Exclusion Criteria:

* Do not speak and understand Danish sufficiently to fill out questionnaires (due to dementia, some foreigners etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with care pathways(questionnaire) | 8, 30 and 52 weeks after inclusion and randomization
Quality of Life measures(questionnaire) | 8, 30 and 52 weeks after inclusion and randomization

SECONDARY OUTCOMES:
Use of health care services during "the secondary care treatment period", i.e. GPs, emergency department, planned and emergency admission, total length of hospitalisation | 12 (and 6) months from diagnosis
GPs' evaluations of continuity of care (questionnaire). | 30 weeks after the patient's inclusion in the trial
Care process measures in terms of monitoring of data from the National Patient Registry | 12 (and 6) months after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Christian N Wulff, MD, Principal Investigator — Research Unit of General Practice, Odense
Locations (1):
- Department P, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Wulff CN, Vedsted P, Sondergaard J. A randomised controlled trial of hospital-based case management to improve colorectal cancer patients' health-related quality of life and evaluations of care. BMJ Open. 2012 Nov 21;2(6):e001481. doi: 10.1136/bmjopen-2012-001481. Print 2012. PMID 23175735